CLINICAL TRIAL: NCT00782561
Title: A Phase I, Open-Label Study of the Safety and Pharmacokinetics of FG-3019 in Adolescent and Adult Subjects With Steroid-Resistant Focal Segmental Glomerulosclerosis
Brief Title: Safety and Pharmacokinetics of FG-3019 in Adolescents and Adults With Focal Segmental Glomerulosclerosis (FSGS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-MC3019-026
Record Dates: First submitted 2008-10-27; First posted 2008-10-31 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: steroid resistant focal segmental glomerulosclerosis; FSGS; adolescent focal segmental glomerulosclerosis; focal segmental glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — pamrevlumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FG-3019 (Experimental): FG-3019 5 mg/kg
  Interventions: Drug: FG-3019

INTERVENTIONS:
Drug: FG-3019 — FG-3019 5 mg/kg IV given over 2 hours every 2 weeks for 8 weeks

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of FG-3019 administered over 8 weeks to adolescent and adult subjects with steroid-resistant focal segmental glomerulosclerosis (FSGS).

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-64 years, inclusive, and girls age 10-11 years, inclusive if Tanner stage 3 or greater
2. Biopsy diagnosis of primary FSGS with biopsy confirmed centrally
3. Age less than or equal to 2 years old at onset of proteinuria
4. First morning urine protein/creatinine ratio (U p/c) >1 gm/gm
5. Estimated glomerular filtration rate greater than or equal to 40 mL/min/1.73 m2

Exclusion Criteria:

1. Non-FSGS renal disease other than benign cyst; or secondary FSGS
2. History of organ transplantation
3. History of allergic or anaphylactic reaction to human, humanized, chimeric or murine monoclonal antibodies
4. History of malignancy, cardiovascular disease, diabetes mellitus, sickle cell disease, multiple sclerosis, systemic lupus erythematosus, or active or recurrent serious infections (including but not limited to Hepatitis B, Hepatitis C, or HIV)
5. Participation in studies of investigational drugs within 6 weeks prior to Day 0 or receipt of an investigational drug within 12 weeks prior to Day 0
6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times the upper limit of normal
7. Hematocrit < 30%

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2009-06-18 (Actual); Study Completion 2009-06-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of FG-3019 as measured by AEs, SAEs, physical exams, lab tests, and the Treatment Satisfaction Questionnaire for Medications | 32 weeks

SECONDARY OUTCOMES:
Standard plasma and urinary PK parameters | 32 weeks
Change from baseline in urinary protein/creatinine, albumin/creatinine, albumin excretion rate, estimated glomerular filtration rate (eGFR), 24 hour urinary protein and fasting serum lipids | 8 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - New Hyde Park, New York
  - Chapel Hill, North Carolina
  - Columbus, Ohio